CLINICAL TRIAL: NCT07359235
Title: A Clinical Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of Recombinant Oncolytic Adenovirus Injection (KD01) Via Intravesical Instillation in Bladder Cancer (BC)
Brief Title: Safety, Tolerability, and Preliminary Efficacy of KD01 Via Intravesical Instillation in Bladder Cancer (BC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zheng Liu, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-TJ-KD01T02
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer (BC)
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD01 treatment: (Experimental): Monotherapy with KD01 or combination therapy with KD01 plus AK104 for the treatment of bladder cancer.
  Interventions: Drug: KD01(the recombinant oncolytic adenovirus)

INTERVENTIONS:
Drug: KD01(the recombinant oncolytic adenovirus) — Drug： Phase Ia：KD01(3 dose groups: 2.6×10¹¹ VP, 5×10¹¹ VP, and 1×10¹² VP) Phase Ib: KD01(5×10¹¹ VP) with AK104(6 mg/kg, given intravenously every two weeks) Administration： Phase Ia: KD01 will be administered weekly during weeks 1-6, 13-15, 25-27, 37-39, 49-51, 73, 97. If patients present with CIS and/or high-grade Ta at the first efficacy assessment in week 12, KD01 will be administered weekly during weeks 16-18. Phase Ib Cohort A: KD01 for the same treatment duration as Phase Ia. AK104: The initial 6 doses will be administered, and subsequent doses will be continued based on the investigator's assessment of the patient's condition and the patient's willingness. Phase Ib Cohort B: KD01 will be administered weekly during weeks 1-6,with AK104 (3 doses). A transurethral resection of the bladder tumor (TURBT) is recommended 2-4 weeks after the final KD01 dose for residual or suspicious tumors, with subsequent treatment determined by investigators based on imaging results.

SUMMARY:
Recombinant oncolytic adenovirus injection (KD01) is an oncolytic virus product. Its main component is a conditionally replicative recombinant human type 5 adenovirus, where part of the E3 region has been replaced with the gene encoding the tBid apoptotic protein.AK104 is a humanized bispecific antibody co-targeting PD-1 (Programmed Cell Death Protein 1) and CTLA-4 (Cytotoxic T-Lymphocyte-Associated Antigen 4)-two key immune checkpoint receptors. It is designed as a novel tetrameric construct that preferentially binds to tumor-infiltrating lymphocytes (TILs) co-expressing PD-1 and CTLA-4 in the tumor microenvironment (with higher avidity than in peripheral tissues).This is a Phase I clinical study designed to evaluate the safety, tolerability, and preliminary efficacy of intravesical instillation of recombinant oncolytic adenovirus injection (KD01) in patients with bladder cancer.This study consists of Phase Ia and Phase Ib, where Phase Ia is a dose-escalation stage.The Phase Ia will include histopathologically confirmed non-muscle-invasive bladder cancer (NMIBC) patients with high-risk stratification (including extremely high-risk).The Phase Ib study will include two independent cohorts: Cohort A comprises high-risk non-muscle-invasive bladder cancer (NMIBC) patients (carcinoma in situ [CIS], with or without Ta/T1 stage lesions) who have shown no response to BCG. Cohort B will include T2-4aN0-1M0 stage bladder cancer patients (clinically localized muscle-invasive bladder urothelial carcinoma).

ELIGIBILITY:
Inclusion Criteria:

* 1.The Phase Ia will include histopathologically confirmed non-muscle-invasive bladder cancer (NMIBC) patients with high-risk stratification (including extremely high-risk). High-risk stratification criteria are defined as G3/high-grade tumors that meet any of the following criteria: carcinoma in situ (CIS); stage T1; diameter>3 cm; multiple tumors; or recurrent tumors. The Phase Ib Cohort A will include BCG unresponsive NMIBC patients with carcinoma in situ [CIS], with or without Ta/T1 stage lesions, while Cohort B will include histopathologically confirmed muscle-invasive bladder cancer (cT2-4aN0-1M0).Note: BCG non-response is defined as meeting any of the following criteria: 1. Persistent or recurrent CIS within 12 months after completing adequate BCG treatment; 2. Recurrence of high-grade Ta/Tl disease within 6 months after completing adequate BCG treatment; 3. High-grade T1 disease at first evaluation after induction BCG treatment. (Adequate BCG treatment is defined as: Complete at least 5 out of 6 doses in the initial induction course. plus 2 out of 6 doses from the second induction course, or 2 doses from the 3-dose maintenance course.)
* 2.Excluding Phase Ib Cohort B, participants must either be medically ineligible for radical cystectomy as determined by urologists or have declined the procedure.
* 3.Age 18 to 75 (including 18 and 75).
* 4.Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 1.
* 5.Estimated survival time is ≥2 years.6.No dysfunction of major organs, including but not limited to hematopoietic function and cardiac, pulmonary,hepatic and renal function.

Hematologic system (no history of blood transfusion or hematopoietic growth factor treatment within 14 days)

1. Absolute neutrophil count (ANC)≥1.5×109/L
2. Platelets （PLT）≥75×109/L
3. Hemoglobin （Hb）≥90g/L

Hepatic function

1. Total bilirubin (TBIL)≤1.5× upper limit (ULN)
2. Alanine aminotransferase (ALT)≤3×ULN
3. Aspartate aminotransferase (AST)≤3×ULN

Renal function

1. Creatinine （Cr）≤1.5×ULN
2. Creatinine clearance (Ccr) (Calculation required only if creatinine exceeds 1.5×ULN)>50 mL/min (calculated using the Cockcroft-Gault formula)

Coagulation function

1. Activated Partial Thromboplastin Time (APTT)≤1.5×ULN
2. International normalized ratio (INR)≤1.5×ULN

   * 7.Premenopausal patients must have a negative blood pregnancy test during the screening period;they must agree to use reliable contraceptive methods (barrier contraceptive method or abstinence) with their partners during the trial and for at least 6 months after the last dose.
   * 8.Patients must provide informed consent to the trial and voluntarily sign of a written informed consent form before participating in the trial.

Exclusion Criteria:

* 1.Evidence of metastatic disease, or multiple regional lymph node positivity in the true pelvis, or common iliac lymph node positivity at the screening visit. Accompanied by hydronephrosis.
* 2.Received pelvic external beam radiation therapy within 5 years.
* 3.Prior treatment with adenovirus-based therapies (e.g., oncolytic adenovirus, CanSino's Ad5-nCoV COVID-19 vaccine).
* 4.Symptomatic urinary tract infection or bacterial cystitis (patients can enter the study once the treatment is satisfactory).
* 5.Clinically significant and unexplained elevation of liver or kidney function markers.
* 6.Women who are pregnant or breastfeeding or refuse to use contraception at any time during the study; male patients who are unwilling to use effective contraception.
* 7.A history of malignancy in another organ system in the past 5 years, which the investigator believes may interfere with the conduct of the study or requires systemic study treatment for the malignancy.
* 8.Patients who cannot tolerate intravesical instillation for 1 hour or bladder surgery.
* 9.In addition to immediate postoperative instillation after TURBT , patients who have received anti-tumor treatments (including chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc.) within 4 weeks before the first study drug administration must be excluded. Specifically, patients who have used nitrosourea drugs or mitomycin C within 6 weeks prior to the initial study drug administration must be excluded Patients who have used oral fluorouracil and small-molecule targeted drugs within 2 weeks prior to the first administration of the study drug or within 5 half-lives of the drugs (whichever is longer) must be excluded. Patients who have used TCMs with anti-tumor indications within 2 weeks prior to the first administration must be excluded.
* 10.History of severe cardiovascular and cerebrovascular diseases, including but not limited to:

  1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, or second-to third-degree atrioventricular block;
  2. At rest, the QTcF (calculated from 12-lead ECG) is ≥460ms.
  3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before the first administration;
  4. Patients with NYHA class ≥II or left ventricular ejection fraction (LVEF) <50%, or those with structural heart disease deemed high-risk by other researchers.
  5. Hypertension that is not clinically controlled.
* 11.Patients with autoimmune diseases, or immune system dysfunction, or after organ transplantation.
* 12.Patients with active infection, or those requiring systemic anti-infective therapy (routine prophylactic anti-infective therapy at the clinical trial site is excluded), or those with unexplained fever > 38.5℃ during screening.
* 13.Patients with positive HIV antibodies (HIV-Ab) or Treponema pallidum antibodies; those with active hepatitis B (HBsAg-positive with HBV-DNA>500 IU/ml or above the clinical trial institution's lower limit of detection [only if the lower limit of detection exceeds 500 IU/ml]); and those with active hepatitis C (HCV-positive but HCV-RNA below the clinical trial institution's lower limit of detection are eligible). Patients receiving prophylactic antiviral therapy other than interferon are also eligible.
* 14.Patients with uncontrolled seizures, central nervous system disorders or psychosis with loss of cognitive ability.
* 15.The severity of adverse reactions from prior anti-tumor treatments has not recovered to ≤Level 1 (according to the Common Terminology Criteria for Adverse Events (CTCAE) 5.0), except for toxicities such as hair loss that researchers have determined to be non-safety risks.
* 16.Antiviral therapy is currently required, or antiviral drugs were used within 2 weeks before the first use of the trial drug.
* 17.Participants who received any live virus vaccine for infectious disease prevention within 4 weeks prior to the study drug administration. Examples of live vaccines include, but are not limited to: measles, mumps, rubella, chickenpox/herpes zoster (varicella), yellow fever, rabies, BCG, and typhoid vaccines. Influenza vaccines for injection are generally inactivated virus vaccines and are permitted; however, intranasal influenza vaccines (e.g., FluMisT®) are live attenuated vaccines and are not permitted.
* 18.Patients who have received systemic glucocorticoids (prednisone>10mg or equivalent doses of similar drugs) or other immunosuppressants within 14 days prior to trial drug administration must be excluded. Exceptions include: topical, ocular, intra-articular, intranasal, or inhaled glucocorticoid treatments; and short-term prophylactic glucocorticoid use (e.g., for preventing contrast agent allergies).
* 19.Patients with severe allergy history or allergic constitution.
* 20.Patients with a history of allogeneic hematopoietic stem cell transplantation or organ transplantation must be excluded.
* 21.Other circumstances that the investigator deems inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
SAEs and AEs（Phase Ia） | 2 years
  The incidence of serious adverse events (SAEs), the incidence and severity of adverse events (AEs).
MTD | 2 years
  Phase Ia: The maximum tolerated dose (MTD) is determined based on the incidence of dose-limiting toxicity (DLT).
SAEs and AEs（Phase Ib） | 2 years
  The incidence of serious adverse events (SAEs), the incidence and severity of adverse events (AEs).

SECONDARY OUTCOMES:
CRR(Phase Ia and Phase Ib Cohort A) | 24 months
  Phase Ia and Phase Ib Cohort A: Complete Response (CR) rates at any time points and at 3, 6, 12,15,18, and 24 months.
DOR（Phase Ia and Phase Ib Cohort A） | 24 months
  Phase Ia and Phase Ib Cohort A: Duration of Response (DOR) at these time points.
CRR(Phase Ib Cohort B) | 24 months
  Phase Ib Cohort B: includes the incidence of pathological complete response (pT0N0) .
PRR(Phase Ib Cohort B) | 24 months
  Phase Ib Cohort B: includes the incidence of pathological partial response（<pT2N0）.
Incidence of cystectomy | 24 months
  Incidence of cystectomy during the study.
RFS | 12 months
  The time interval from the completion of curative treatment to the first recurrence of the disease。
Biodistribution | 2 years
  The detected concentrations of KD01 in blood, urine, feces, and saliva in Phase Ia patients.

OTHER OUTCOMES:
Antibodie | 2 years
  Dynamic changes in anti-Ad5 adenovirus antibodies.
Neutralizing antibodies | 2 years
  Dynamic changes in neutralizing antibodies.
Immunogenicity | 2 years
  The immunogenicity of KD01 via ELISPOT or ICS.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China